CLINICAL TRIAL: NCT01820052
Title: A Double-blind , Randomized, Placebo-controlled Trial of Oral Iron Therapy in Fibromyalgia
Brief Title: A Randomized Trial of Oral Iron Therapy in Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-03-DM-67
Record Dates: First submitted 2013-03-21; First posted 2013-03-28 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Primary Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Iron; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Iron (Active Comparator): Patient will receive 230 mg of oral elemental iron daily for 3 months
  Interventions: Drug: Oral Iron
- Oral Placebo (Placebo Comparator): Oral Placebo tablets will be administered daily for 3 months
  Interventions: Drug: Oral Placebo

INTERVENTIONS:
Drug: Oral Iron — 230 mg of elemental oral iron tablets will be administered daily for 3 months
  Other Names: Drug
  Arms: Oral Iron
Drug: Oral Placebo — Oral tablets matching oral iron will be administered daily for 3 months
  Other Names: Placebo
  Arms: Oral Placebo

SUMMARY:
Fibromyalgia (FM) is a disorder with chronic widespread musculoskeletal pain for which no alternative cause can be identified. The condition is often accompanied by other features such as fatigue, stiffness, cold intolerance, cognitive impairment, intolerance to external stimuli, sleep disturbances, anxiety and depression, which significantly affect the quality of life. Fibromyalgia is characterized by altered pain perception, and studies have shown fibromyalgia to be more prevalent in patients with iron deficiency anemia. Iron is essential for a number of enzymes involved in serotonin and dopamine synthesis. Deficiency of serotonergic neuronal functioning might be related to the pathophysiology of FM.

This study attempts to explore the use of oral iron as a cheap and readily available alternative for the treatment of FM .

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a disorder with chronic widespread musculoskeletal pain for which no alternative cause can be identified . The condition is often accompanied by other features such as fatigue, stiffness, cold intolerance, cognitive impairment, intolerance to external stimuli, sleep disturbances, anxiety and depression, which significantly affect the quality of life. Fibromyalgia is characterized by altered pain perception, and studies have shown fibromyalgia to be more prevalent in patients with iron deficiency anemia. Iron is essential for a number of enzymes involved in serotonin and dopamine synthesis. Deficiency of serotonergic neuronal functioning might be related to the pathophysiology of FM. A dysregulation of dopaminergic transmission in the pathophysiology of FM has also been suggested. This has brought forth the postulation that iron as a cofactor in serotonin and dopamine production may have a role in the etiology of FM.

A number of therapies are currently in vogue for FM, both pharmacological and non-pharmacological. Drugs shown to be effective in FM include tricyclic antidepressants(amitryptiline, cyclobenzaprine), dual reuptake inhibitors (duloxetine, milnacipran) and alpha-2-delta ligands (pregabalin, gabapentin). However cost is a major factor, and often treatment results are disappointing . Hence the investigators planned to conduct a randomized controlled trial of iron therapy in fibromyalgia . IF proven, iron could be a cheap and easily available alternative for the treatment of this common and often disabling condition.

Materials and methods:

Patients with FM attending the OPD of the Department of Clinical Immunology will be identified . Diagnosis shall be made as per the ACR 2010 preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. After seeking informed consent, the subjects will undergo baseline investigation to look for Hb, thyroid function tests and 25-OH-Vitamin. Patients with a Hb<8 g or having hypothyroidism , deficiency of Vitamin D or any connective tissue disease will be excluded from the study. Patients with a baseline FIQ >40 will be taken up for study. Baseline depression will be assessed using BPHQ and patients with a baseline BPHQ > 4 will be excluded from study. Following this, the patients will undergo assessment of serum ferritin at baseline, and irrespective of serum ferritin levels, will be randomized into 2 groups. Target sample size in each group will be 60. The groups will be blinded from both the patients and the investigators, and allocation concealment will be maintained by use of pre-sealed envelopes and drug packets. Group A will receive standard of care treatment for fibromyalgia (Amitryptiline up to 25 mg/day, Duloxetine upto 60 mg/day, Pregabalin upto 300 mg/day either singly or in combination) along with placebo for 3 months. Group B will receive standard of care treatment for fibromyalgia (Amitryptiline upto 25 mg/day, Duloxetine upto 60 mg/day, Pregabalin up to 300 mg/day either singly or in combination) along with 230 mg of oral elemental iron daily for 3 months. Assessment at baseline and at 3 months will be done with respect to the primary end points - Widespread Pain Index (WPI), Symptom Severity Scale score (SSS), Hindi version of Fibromyalgia Impact Questionnaire (FIQ) , and secondary end points - Visual Analog Scale for pain (VAS) , Hindi version of Brief Physical Health Questionnaire (BPHQ) , Hindi version of SF-36 questionnaire. Patients will be monitored for side effects of oral iron therapy ( nausea,vomiting, gastrointestinal irritation , constipation , diarrhea) . At the end of 3 months, statistical analysis will be done to determine significance of difference between placebo groups A and B with respect to the above mentioned end points. Patients with a change in FIQ > 25% will be taken as responders. The change in levels of various end points before and after, viz. WPI, SSS, VAS, BPHQ, SF-36 will be a secondary consideration.

Significance:

This study attempts to explore the use of oral iron as a cheap and readily available alternative for the treatment of FM .

ELIGIBILITY:
Inclusion Criteria:

* Patients of Fibromyalgia fulfilling ACR 2010 criteria.
* Patients with a baseline FIQ >40 will be taken up for study.

Exclusion Criteria:

* Patients with a Hb<8 g or having hypothyroidism , deficiency of Vitamin D or any connective tissue disease will be excluded from the study.
* Baseline depression will be assessed using BPHQ and patients with a baseline BPHQ > 4 will be excluded from study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Widespread Pain Index | Change from baseline to 3 months
  Patient reported Widespread Pain Index (WPI)
Symptom Severity Scale score | Change from baseline to 3 months
  Patient reported Symptom Severity Scale score
Hindi version of Fibromyalgia Impact Questionnaire | Change from baseline to 3 months
  Patient reported Hindi version of Fibromyalgia Impact Questionnaire

SECONDARY OUTCOMES:
Visual Analog Scale for pain | Change from baseline to 3 months
  Patient reported Visual Analog Scale for pain on a 10 cm scale
Hindi version of Brief Physical Health Questionnaire | Change from baseline to 3 months
  Patient reported Hindi version of Brief Physical Health Questionnaire
Hindi version of SF-36 questionnaire. | Change from baseline to 3 months
  Patient reported Hindi version of SF-36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Agarwal, MD, DM, Principal Investigator — Additional Professor, Clinical Immunology
Locations (1):
- SGPGIMS, Lucknow, Uttar Pradesh, India